CLINICAL TRIAL: NCT02749409
Title: Early Parecoxib Usage to Decreases Narcotic Requirement and Length of Stay After Traumatic Rib Fracture
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Case numbers not enough, however, the funding is over
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARECOXIB RIB
Record Dates: First submitted 2016-04-07; First posted 2016-04-25 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2016-07

CONDITIONS: Parecoxib; Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — parecoxib; Morphine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control group (Active Comparator): The control group will be given Morphine prn after admission
  Interventions: Drug: Morphine
- Experimental group (Experimental): the experimental group will be given parecoxib after admission by intravenous method every 12 hours for 4 days. Then Morphine agent will be given prn usage
  Interventions: Drug: Parecoxib

INTERVENTIONS:
Drug: Parecoxib
  Arms: Experimental group
Drug: Morphine
  Arms: Control group

SUMMARY:
Patients diagnosed traumatic rib fracture and need admission will be included. Patients will be divided two groups.The experimental group will be given parecoxib after visiting emergency department. The control group will be given Narcotic agent such as morphine for pain control. The outcome such as numerical rating scale (NRS) and hospital length of stay will be recorded.

DETAILED DESCRIPTION:
3.1 Inclusion/exclusion criteria Patients who are diagnosed ribs fracture and need admission. Exclusion criteria included heart failure, Coronary artery disease (CAD) history. Traumatic cardiac injury and cardiac tamponade will be excluded, too.

3.2 Group design Patients will be divided two groups, and the experimental group will be given parecoxib after visiting emergency department. And they will be kept given after admission by intravenous method every 12 hours for 4 days. The control group will be given Narcotic agent such as morphine for pain control. The daily dose will be recorded. Finally the end outcome will be recorded.

3.3 Data collection The data of patient's medical history and laboratory results will be recorded on pre-designed case report forms (CRFs) by study nurses. In all patients, age, gender, diagnosis, co-morbidities, length of hospital and intensive care unit (ICU) stay, Injury Severity Score (ISS) score, numerical rating scale (NRS) and outcomes, will be recorded. In addition, all microorganisms isolated and antibiotic substances applied will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Investigators will prospective enroll patients who are diagnosed chest trauma with rib fractures
2. Age ≧18 y/o

Exclusion Criteria:

1. Patients who have history of heart failure, CAD history.
2. Traumatic cardiac injury and cardiac tamponade
3. History of allergy effect for Cyclooxygenase 2 (COX2) inhibitor or NSAID

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 1 year